CLINICAL TRIAL: NCT05327725
Title: Fatigue Reduction Diet in Survivors of Diffuse Large B-Cell Lymphomas; a Preliminary Study
Brief Title: Fatigue Reduction Diet in Lymphoma Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Tonya Orchard, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20182
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Fatigue
Keywords: fatigue reduction diet
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fatigue Reduction Diet Intervention (Experimental): Participants receive individualized nutrition counseling to adopt the fatigue reduction diet protocol via 8 remote phone or video telehealth sessions with a registered dietitian over 3 months.
  Interventions: Other: Fatigue Reduction Diet

INTERVENTIONS:
Other: Fatigue Reduction Diet — Participants receive individualized nutrition counseling to adopt the fatigue reduction diet protocol.

SUMMARY:
The purpose of this small preliminary study is to gather preliminary data to support a large randomized controlled trial of a fatigue reduction diet intervention among diffuse-large B-cell lymphoma (DLBCL) survivors. This study will provide nutritional counseling to 10 adult patients (18 years or older) with DLBCL who have completed their upfront chemotherapy treatment and remained in remission for 2 years prior to enrollment. The study will employ individualized dietary counseling, provided by a registered dietitian (RD), by phone or video teleconferencing in 8 sessions over 3 months. Dietary intake and fatigue will be assessed at baseline and 3 months. The objective of the study is to determine feasibility of the intervention and adherence to the fatigue reduction diet. Data obtained from this preliminary study would be used to support a well-powered future randomized trial of FRD vs regular diet in survivors of DLBCL.

DETAILED DESCRIPTION:
Fatigue is highly prevalent in survivors of diffuse-large B-cell lymphoma (DLBCL). Fatigue has been linked to chronic inflammation, and diets high in antioxidant nutrients (diet rich in fruit, vegetables, whole grains, and omega-3 fatty acid-rich foods) have been associated with lesser prevalence and severity of fatigue. Studies are needed, however, to test if antioxidant-rich diets could improve fatigue in this patient population. This fatigue-reducing diet (FRD) was shown to improve fatigue and sleep in breast cancer survivors compared to regular diet. This FRD diet aligns with the standard of care dietary recommendations for cancer survivors promoted by the American Cancer Society (ACS) . The purpose of this small preliminary study is to gather preliminary data to support a large randomized controlled trial. This study will provide nutritional counseling to 10 adult patients (18 years or older) with DLBCL who have completed their upfront chemotherapy treatment and remained in remission for 2 years prior to enrollment. The study will employ individualized dietary counseling, provided by a registered dietitian (RD), by phone or video teleconferencing. Phone counseling will be weekly for the first month, and then biweekly for the next two months, for a total of 8 phone sessions. Counseling sessions take ~15-30 minutes. Dietary intake will be assessed using an electronic food frequency questionnaire at baseline and 3 months. Fatigue will be assessed using an online survey at baseline and 3 months. The purpose of the study to ascertain the percentage of patients who are able to complete all the study questionnaires and visits and adhere to the fatigue reduction diet. Data obtained from this preliminary study would be used to support a well-powered future randomized trial of FRD vs regular diet in survivors of DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18+) with Diffuse large B-cell lymphoma (DLBCL) who have completed their upfront chemoimmunotherapy, and remained in remission for 2 years prior to enrollment

Exclusion Criteria:

* Unable to provide consent or speak English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | 3 months
  Determine feasibility of recruiting, enrolling and retaining participants in the study, represented as percentage of patients who completed the study.
Adherence to fatigue reduction diet | 3 months
  Determine percentage of patients who adhered to the fatigue reduction diet protocol

CONTACTS AND LOCATIONS:
Overall Officials: Tonya Orchard, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No